CLINICAL TRIAL: NCT05426278
Title: The Effect Of Intraoperative Forced Air Warmer Use, On Postoperative Nausea And Vomiting Among Laparoscopic Surgery Patients: A Randomized Controlled Trial
Brief Title: The Effect Of Intraoperative Forced Air Warmer Use, On Postoperative Nausea And Vomiting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Mohammad Hamid, Associate professor, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2022-7343-21332
Record Dates: First submitted 2022-06-10; First posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Hypothermia; Anesthesia; Nausea and Vomiting, Postoperative
MeSH Terms: conditions — Hypothermia; Postoperative Nausea and Vomiting

STUDY DESIGN:
Intervention Model Description: 2 groups will be made - One group will be interventional and the Other will be the Control group
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FAW and Bair Hugger Group (Other): Group B, the intervention group (with FAW and Bair Hugger).
  Interventions: Device: Bair hugger and Forces air warmer
- Control group (No Intervention): Group A, the control group (No FAW or Bair Hugger)

INTERVENTIONS:
Device: Bair hugger and Forces air warmer — The EQUATOR™ (EQ-5000) air-warmer is a convective warmer, with the average and maximum Contact Surface Temperatures of 39℃ & 44℃ Respectively. Temperature on this device can be set at 36℃ , 40℃ , 44℃. The 3M™ Bair Hugger ™ (SW-2003) upper body blanket is used to warm the body from head till the xiphisternum
  Arms: FAW and Bair Hugger Group

SUMMARY:
Intraoperative Hypothermia is a common problem, our object will be to evaluate the efficacy of forced air warmer (Model # eq-5000) for maintaining core body temperature in patients undergoing laparoscopic surgeries and its effect on postoperative nausea, vomiting and shivering.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing laparoscopic surgeries (Hernia Repair, Cholecystectomy, Appendectomy, Hysterectomy)
* ASA Category I and II as per American Society of Anaesthesiologist Classification.
* BMI< 35 kg/m2
* Duration of surgery >1 hour and <3 hours
* Patients who consent their participation

Exclusion Criteria:

* Temperature >37.5oC or <35oC,
* Chronic kidney disease
* Heart failure
* ASA Category 3&4 (American Society of Anaesthesiologist Classification)
* Patients will be withdrawn from the group if their laparoscopy is converted to open surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Post Operative Nausea Vomiting Scale | Day 1
  The scores of 0-3 will determine severity on the Post-operative nausea and vomiting scale.
  0 - No nausea , No vomiting
  1. - Nausea present , No Vomiting
  2. - Nausea present , Vomiting present
  3. - Vomiting >2 episodes within 30 minutes
Bedside Shivering Assessment Scale (BSAS) | Day 1
  The scores of 0-3 will determine severity on Shivering
  0 -(none) No shivering is detected on palpation of masseter, Neck, or chest muscles
  1. -(mild) Shivering localized to Neck and thorax only
  2. -(moderate) Shivering involves gross movement of the upper extremities( in addition to neck and thorax)
  3. -(severe) Shivering involves gross movements of the trunk and upper and lower extremities

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Torossian A, Brauer A, Hocker J, Bein B, Wulf H, Horn EP. Preventing inadvertent perioperative hypothermia. Dtsch Arztebl Int. 2015 Mar 6;112(10):166-72. doi: 10.3238/arztebl.2015.0166. PMID 25837741
- [Background] Pyzocha NJ, Steele JL. Hypothermia in adults: A strategy for detection and Tx. J Fam Pract. 2018 May;67(5):E1-E7. PMID 29726859
- [Background] Putzu M, Casati A, Berti M, Pagliarini G, Fanelli G. Clinical complications, monitoring and management of perioperative mild hypothermia: anesthesiological features. Acta Biomed. 2007 Dec;78(3):163-9. PMID 18330074
- [Background] Liang D, Shan Y, Wang L. The effect of prophylactic rewarming on postoperative nausea and vomiting among patients undergoing laparoscopic hysterectomy: a prospective randomized clinical study. Sao Paulo Med J. 2020 Sep-Oct;138(5):414-421. doi: 10.1590/1516-3180.2020.0059.R2.06072020. PMID 33053048